CLINICAL TRIAL: NCT05128968
Title: Impact of Head and Neck Positions on Endotracheal Intubation Using a McGRATH MAC Video Laryngoscope
Brief Title: Head and Neck Positions for Endotracheal Intubation Using a Videolaryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Professor, SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 11-2021
Record Dates: First submitted 2021-11-11; First posted 2021-11-22 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Endotracheal Intubation
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Simple extension (Experimental): After induction of anesthesia, endotracheal intubation was performed in simple extension without a pillow using a McGrath MAC videolaryngoscope.
  Interventions: Procedure: endotracheal intubation
- Head elevated position (Experimental): After induction of anesthesia, endotracheal intubation was performed in a head elevated position with a pillow using a McGrath MAC videolaryngoscope.
  Interventions: Procedure: endotracheal intubation
- Sniffing position (Experimental): After induction of anesthesia, endotracheal intubation was performed in a sniffing position using a McGrath MAC videolaryngoscope.
  Interventions: Procedure: endotracheal intubation

INTERVENTIONS:
Procedure: endotracheal intubation — Endotracheal intubation is performed in simple head extension or sniffing position using a McGrath MAC videolaryngoscope.

SUMMARY:
In this study, the investigators evaluate the effect of head positions (simple extension vs. sniffing position vs. head elevation) on endotracheal intubation using a videolaryngoscope.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for general anesthesia

Exclusion Criteria:

* Limited neck extension
* Anatomical anomalies or history of surgery in the upper airway
* Weak teeth
* Risk of pulmonary aspiration

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Ease of intubation | Procedure (During endotracheal intubation)
  Ease of endotracheal intubation is assessed using the intubation difficulty scale.
  Intubation difficulty scale includes number of attempts, number of operators, number of alternative techniques, glottic opening and so on.

SECONDARY OUTCOMES:
Percentage of glottic opening (POGO) score | Procedure (During endotracheal intubation)
  POGO score is recorded during endotracheal intubation (0%: no visualization of glottic opening; 100%: entire visualization of the glottic opening).
Number of attempts | Procedure (At the end of endotracheal intubation)
  Number of attempts for endotracheal intubation is recorded.
Intubation time | Procedure (During endotracheal intubation)
  The time taken for endotracheal intubation is recorded.
Palatopharyngeal wall injury | Procedure (During endotracheal intubation)
  Presence of palatopharyngeal wall injury is observed.
Lifting force for exposure of the glottis | Procedure (During endotracheal intubation)
  Requirement for lifting force to expose the glottis is recorded during videolaryngoscopy
Laryngeal pressure for exposure of the glottis | Procedure (During endotracheal intubation)
  Requirement for laryngeal force to expose the glottis is recorded during videolaryngoscopy
Lifting force for advancing an endotracheal tube into the larynx | Procedure (During endotracheal intubation)
  Requirement for lifting force is recorded during the advancement of the endotracheal tube into the larynx.
Laryngeal pressure for advancing an endotracheal tube into the larynx. | Procedure (During endotracheal intubation)
  Requirement for laryngeal pressure is recorded during the advancement of the endotracheal tube into the larynx.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Young Hwang, PhD., Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim H, Chang JE, Won D, Lee JM, Kim TK, Kim MJ, Min SW, Hwang JY. Effect of head and neck positions on tracheal intubation using a McGRATH MAC video laryngoscope: A randomised, prospective study. Eur J Anaesthesiol. 2023 Aug 1;40(8):560-567. doi: 10.1097/EJA.0000000000001838. Epub 2023 Apr 13. PMID 37052067